CLINICAL TRIAL: NCT04769128
Title: INFLUENCE of THORACIC MANIPULATION on TYPE 1 COMPLEX REGIONAL PAIN SYNDROME Post-UPPER LIMB TRAUMA
Brief Title: THORACIC MANIPULATION and COMPLEX REGIONAL PAIN SYNDROME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Manal Mohammed Hassan, principal investigator, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Thoracic manipulation on CRPS1
Record Dates: First submitted 2021-02-20; First posted 2021-02-24 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (control group)(traditional physical therapy programme) (Active Comparator): Group (A) (control group): Fifteen patients with CRPS I received traditional physical therapy program in the form of transcutaneous electrical neuromuscular stimulation (TENS), mirror therapy, and exercises for upper limb exercises in the form of gradual weight-bearing exercises by using different equipment such as balls, balloons, or silk-like cloths, combined with different positions of the patient (i.e. lying, sitting, or standing), range of motion exercises (active and self-Assisted), resisting exercises (manual and mechanical), stretching exercises (manual and self-stretching) and fine motor control training. 3 sessions/ week for 12 weeks.
  Interventions: Other: Traditional physical therapy programe
- Group (B) (experimental or manipulative group) (Experimental): Fifteen patients with CRPS I received traditional physical therapy program in the form of transcutaneous electrical neuromuscular stimulation (TENS), mirror therapy, and exercises for upper limb exercises in the form of gradual weight-bearing exercises by using different equipment such as balls, balloons, or silk-like cloths, combined with different positions of the patient (i.e. lying, sitting, or standing), range of motion exercises (active and self-Assisted), resisting exercises (manual and mechanical), stretching exercises (manual and self-stretching) and fine motor control training in addition to T3-T4 thoracic manipulation (Maitland "screw" technique grade V) 3 sessions/ week for 12 weeks.
  Interventions: Other: Traditional physical therapy programe

INTERVENTIONS:
Other: Traditional physical therapy programe — thoracic manipulation spine at the level of T3 and T4 facet joints (Maitland (screw) technique grade V). Using hypothenar eminence of hands, applying direct downward pressure and additional force-directed caudal with one hand and cephalic with the other hand on the transverse processes.
  Other Names: Thoracic manipulation

SUMMARY:
To compare the effect of combined thoracic manipulation (TM) and traditional physical therapy treatment (TPT) versus TPT treatment alone on pain severity at rest and functional disability in patients with type 1 complex regional pain syndrome (CRPS I) post-upper limb trauma.

DETAILED DESCRIPTION:
Complex regional pain syndrome (CRPS) is a chronic state of pain that is frequently triggered by an injury and is characterized by a variable combination of sensory, motor, vasomotor, and sudomotor symptoms, in the affected limb..the frequency of CRPS after injury was 3.8-7.0 % within four months of fracture. The highest prevalence occurs in the age group of 40 to 60 years. The pathophysiology of CRPS is still controversial, but a recent study has shown that up to 70% of patients with CRPS have anti-autonomic immunoglobulin G (IgG) autoantibodies associated with autonomic disorders in their serum CRPS, increasing the probability of these antiautonomic antibodies contributing to the pathophysiology of CRPS. Under normal conditions, sympathetic behavior does not affect the discharge of nociceptors; but nociceptors tend to be under the control of the sympathetic nervous system (SNS) in the case of CRPS. This is referred to as pain maintained sympathetically. Conservative treatments for CRPS I have traditionally focused on pain reduction through pharmacology, desensitization therapy, transcutaneous electrical stimulation (TENS), and thermal modalities and function restoration through active, passive, and strengthening exercises of the arm.

Patients with arm CRPSI also show postural deviations related to the arm's defensive role. During all upright tasks, this posture reduces trunk motion and can have effects such as reduced thoracic intervertebral mobility. Near to the thoracic costovertebral and zygapophyseal joints are the sympathetic chain ganglia that innervate the upper limb. It may be probable that the sympathetic chain ganglia affected by thoracic dysfunction arising from joint or soft tissue restriction and may be related to the distal symptoms in CRPS. Thus, thoracic spine manipulation can be an aid to the overall treatment of the symptoms in patients with CRPS I. There is no study involving a control group in the available studies. As with all case studies, while the findings might be interesting for future research. our study is the first study to investigate the impact of thoracic manipulation in patients with CRPS1 by comparing between the control group and the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Thirty patients were diagnosed according to International Association for the Study of Pain (IASP) criteria with CRPS I (10 to 18 weeks duration of illness) from both genders and referred from orthopedists post fractures in different upper limb regions (such as shoulder region e.g. clavicle and proximal humerus, elbow region e.g. distal humerus, proximal radius and ulna, and wrist region e.g. distal radius, ulna, and carpal bones), their age was between 40 and 60 years.

Exclusion Criteria:

* Patients who had a stroke, any history of autoimmune or peripheral vascular diseases, diabetes, T4 syndrome, as well as patients, received physical therapy program before

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-29 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
analog scale (VAS) | during 1 day
  The patient is asked to draw a line at the point that represents their pain severity perpendicular to the VAS line. The score is measured by calculating the distance (mm) on the 10-cm line between the 'no pain' anchor and the mark of the patient by using a ruler, including a selection of scores from 0-100. A higher score indicates greater pain intensity. The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44mm), moderate pain (45-74 mm), and severe pain (75- 100 mm). A difference of more than 12 mm is considered the minimum clinically important difference. The patient rated the pain severity at rest.
functional disability using disability of arm, shoulder, and hand questionnaire (DASH). | 1 week
  DASH is a self-assessment of symptoms and function of the entire upper extremity. Self-assessment and scoring by calculating the arithmetic mean of at least 27 of the 30 items (missing rule) is transformed by (mean - 1) x 25 into the scale from 0 no symptoms/full function to 100 maximal symptoms/no function for the DASH total score. Five of 6 items are necessary for determination of the symptoms score and 22 of 24 items for the function score. Originally, 0 best and 100 worst. All items are easy to comprehend and are not emotionally sensitive (with the exception of item 21). All items are scored on a scale of 5 (Likert) levels: (1) no difficulty/ symptoms, (2) mild difficulty/ symptoms, (3) moderate difficulty/symptoms, (4) severe difficulty/ symptoms, and (5) extreme difficulty (unable to do)/symptoms. Minimal Clinical Important Difference (MCID): 10.2 points. In our current study, the Arabic version was used

CONTACTS AND LOCATIONS:
Overall Officials: Manal M Hassan, Msc, Principal Investigator — out pateints clinic, faculty of physical therapy, SVU, Qena. Eygpt. info@pt.svu.edu.eg. 201061792003
Locations (1):
- Manal M Hassan, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marinus J, Moseley GL, Birklein F, Baron R, Maihofner C, Kingery WS, van Hilten JJ. Clinical features and pathophysiology of complex regional pain syndrome. Lancet Neurol. 2011 Jul;10(7):637-48. doi: 10.1016/S1474-4422(11)70106-5. PMID 21683929
- [Result] Beerthuizen A, Stronks DL, Van't Spijker A, Yaksh A, Hanraets BM, Klein J, Huygen FJPM. Demographic and medical parameters in the development of complex regional pain syndrome type 1 (CRPS1): prospective study on 596 patients with a fracture. Pain. 2012 Jun;153(6):1187-1192. doi: 10.1016/j.pain.2012.01.026. Epub 2012 Mar 3. PMID 22386473
- [Result] Bruehl S, Maihofner C, Stanton-Hicks M, Perez RS, Vatine JJ, Brunner F, Birklein F, Schlereth T, Mackey S, Mailis-Gagnon A, Livshitz A, Harden RN. Complex regional pain syndrome: evidence for warm and cold subtypes in a large prospective clinical sample. Pain. 2016 Aug;157(8):1674-81. doi: 10.1097/j.pain.0000000000000569. PMID 27023422
- [Result] Kohr D, Singh P, Tschernatsch M, Kaps M, Pouokam E, Diener M, Kummer W, Birklein F, Vincent A, Goebel A, Wallukat G, Blaes F. Autoimmunity against the beta2 adrenergic receptor and muscarinic-2 receptor in complex regional pain syndrome. Pain. 2011 Dec;152(12):2690-2700. doi: 10.1016/j.pain.2011.06.012. Epub 2011 Aug 3. PMID 21816540
- [Result] Dubuis E, Thompson V, Leite MI, Blaes F, Maihofner C, Greensmith D, Vincent A, Shenker N, Kuttikat A, Leuwer M, Goebel A. Longstanding complex regional pain syndrome is associated with activating autoantibodies against alpha-1a adrenoceptors. Pain. 2014 Nov;155(11):2408-17. doi: 10.1016/j.pain.2014.09.022. Epub 2014 Sep 22. PMID 25250722
- [Result] Sillevis R, Cleland J, Hellman M, Beekhuizen K. Immediate effects of a thoracic spine thrust manipulation on the autonomic nervous system: a randomized clinical trial. J Man Manip Ther. 2010 Dec;18(4):181-90. doi: 10.1179/106698110X12804993427126. PMID 22131791
- [Result] Benarroch EE. Pain-autonomic interactions. Neurol Sci. 2006 May;27 Suppl 2:S130-3. doi: 10.1007/s10072-006-0587-x. PMID 16688616
- [Result] Vernon HT, Triano JJ, Ross JK, Tran SK, Soave DM, Dinulos MD. Validation of a novel sham cervical manipulation procedure. Spine J. 2012 Nov;12(11):1021-8. doi: 10.1016/j.spinee.2012.10.009. Epub 2012 Nov 15. PMID 23158966
- [Result] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Result] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Result] Angst F, Goldhahn J, Drerup S, Flury M, Schwyzer HK, Simmen BR. How sharp is the short QuickDASH? A refined content and validity analysis of the short form of the disabilities of the shoulder, arm and hand questionnaire in the strata of symptoms and function and specific joint conditions. Qual Life Res. 2009 Oct;18(8):1043-51. doi: 10.1007/s11136-009-9529-4. Epub 2009 Aug 26. PMID 19707887
- [Result] Packham T, Holly J. Complex regional pain syndrome: Measurement matters: Re: Galve-Villa M, Rittig-Rasmussen B, Mikkelsen LMS, Poulsen AG. Complex Regional Pain Syndrome. Manual Therapy 2016;26:e2-3. Man Ther. 2016 Dec;26:e1. doi: 10.1016/j.math.2016.07.012. Epub 2016 Aug 2. No abstract available. PMID 27527554
- [Result] Harden RN, Oaklander AL, Burton AW, Perez RS, Richardson K, Swan M, Barthel J, Costa B, Graciosa JR, Bruehl S; Reflex Sympathetic Dystrophy Syndrome Association. Complex regional pain syndrome: practical diagnostic and treatment guidelines, 4th edition. Pain Med. 2013 Feb;14(2):180-229. doi: 10.1111/pme.12033. Epub 2013 Jan 17. PMID 23331950